CLINICAL TRIAL: NCT03812614
Title: Comparative Effectiveness of Adding Family Supporter Training to a CHW-Led Intervention to Improve Behavioral Management of Multiple Risk Factors for Diabetes Complications
Brief Title: Comparative Effectiveness of Family vs. Individually Focused Diabetes Education and Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Community Health and Social Services Center, Inc. (Other); University of Michigan (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ann-Marie Rosland, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY20110344; R01DK116733 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; High Blood Pressure; High Blood Sugar; Hypertension
Keywords: Diabetes; Patient Activation; Self Management Education; Self Management Behavior; Autonomy Support; Social Support; Caregiver; Family Support; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperglycemia; Patient Participation | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This is a randomized comparative effectiveness trial comparing two interventions.
  The participants and staff delivering the interventions will not be blinded, but the data analyst will be.
  This trial aims to compare the effect of the FAM-ACT intervention on patients' diabetes-related health behaviors and outcomes compared to patient-focused DSME and support (I-DSMES).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes Assessor will be unaware of the arm assignment of the participant when assessing main outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAM-ACT (Experimental): Patient and Support Person (dyad) will be included together as much as possible. The dyad will:
  1. Take part in a one-hour introductory session and review of the patient's Diabetes Complications Risk Assessment profile.
  2. Be invited to 4-6 Support Person-focused, group diabetes self-management education (DSME) sessions lasting 1-2 ½ hours each.
  3. Receive case management contacts with a Community Health Worker (CHW) once every 2-4 weeks, subject to participant availability. Successful contacts will last approximately 20 minutes.
  Interventions: Behavioral: FAM ACT
- I-DSMES (Active Comparator): This arm will focus on the patient only. The Support Person assigned to this arm will not be invited to the introduction sessions, care management contacts, or diabetes self-management education sessions. Patients assigned to this arm will:
  1. Take part in a one-hour introductory session and review of patient's diabetes management risk assessment.
  2. Be invited to 4-6 group diabetes self-management education (DSME) sessions lasting 45 min to 2 hours each.
  3. Receive case management contacts with a Community Health Worker (CHW) once every 2-4 weeks, subject to participant availability. Successful contacts will last approximately 20 minutes.
  Interventions: Behavioral: I-DSMES

INTERVENTIONS:
Behavioral: FAM ACT — Patient and Support Person (dyad) will receive a Diabetes Complications Risk Assessment profile and introduction session, Support Person-focused information/skills training through 4-6 extended DSME sessions, case management contacts with CHW throughout the duration of the 6-month intervention, and guidance on how to prepare for and participate in healthcare appointments.
  Other Names: Family Support for Health Action
  Arms: FAM-ACT
Behavioral: I-DSMES — Patient only will receive a Diabetes Complications Risk Assessment profile and introduction session, 4-6 group DSME sessions, case management contacts with CHW throughout the duration of the 6-month intervention, and guidance on how to prepare for and participate in healthcare appointments.
  Other Names: Individual-Focused DM Self-Management Education and Support
  Arms: I-DSMES

SUMMARY:
The objective of this study is to compare the effectiveness of a novel program-Family Support for Health Action (FAM-ACT) - to individual patient-focused diabetes self-management education and support (I-DSMES).

DETAILED DESCRIPTION:
FAM-ACT uses three innovative approaches to enhance the impact of family support on diabetes management for adults with diabetes (AWDs):

1. coach family supporters in regular discussions about AWDs' diabetes progress and goals that uses empathetic and autonomy-supportive communication,
2. coach family supporters in practical roles that support diabetes-specific tasks tailored to AWDs' personal goals,
3. leverage family support in the setting of other types of social support for AWDs (support from other AWDs and their family members and Community Health Workers (CHWs))

FAM-ACT will be developed and implemented in culturally-concordant ways, in partnership with the community participating in the program.

Adults with type 2 diabetes and either poor glycemic or blood pressure control will be randomized together with a Support Person (a chosen adult family member or friend) to receive either FAM-ACT or more traditional CHW-led patient-focused I-DSMES over 6 months.

See our published protocol (Deverts et al 2022; full citation in references section) for additional details on the protocol including any changes made after the study started.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Have a diagnosis of Type 2 diabetes
2. Most recent HbA1c done in the 3 months prior to screening phone call >= 7.5%
3. Plan to use recruiting site for health care over the next 12 months after enrollment
4. Must be able to identify a family member or friend who is willing to be involved in their health care

Patient Exclusion Criteria:

1. Diagnosis (active or prior) of Alzheimer's disease or dementia
2. Preferred language is not English or Spanish
3. Diagnosis (active or prior) of schizophrenia or other psychotic/delusional disorder in CHASS EMR Problem list as of screening call date
4. Diagnosis of gestational diabetes without any other diabetes diagnoses
5. Diagnosed with diabetes at age < 21 years
6. Pregnant or planning to become pregnant in the next 12 months
7. Concerns that may make it difficult to participate (ongoing health issues, personal events, etc.)
8. Have a life-limiting severe illness (e.g. chronic obstructive pulmonary disease requiring oxygen)

Support Person Inclusion Criteria:

1. Able to attend intervention sessions in person or remotely via online video-conferencing
2. At least 21 years old

Support Person Exclusion Criteria:

1. Does not speak English or Spanish
2. Receives pay for caring for the patient
3. Has self-reported serious mental illness (schizophrenia)
4. Has a life-limiting severe illness (e.g. chronic obstructive pulmonary disease requiring oxygen)
5. Has significant cognitive impairment (Alzheimer's disease or dementia)
6. Lives in a nursing home or long-term care facility
7. Concerns that may make it difficult to participate (ongoing health issues, personal events, etc.)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie Rosland, MD,MS, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Community Health and Social Services Center (CHASS), Detroit, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The study investigators will make de-identified data sets available for sharing after the trial is finished and primary analyses have been completed and published. Researchers requesting data must present an IRB-approved methodological protocol and explain the relevance of their interest in the study completed data to public health goals. Authors completing secondary analyses of the shared study data must agree to the Center for Clinical Trials and Data Coordination (CCDC) policy on data sharing and publishing. All secondary analysis authors will be expected to credit the primary investigators and mention the data source in all publications. Secondary authors will acknowledge that the data use was in accordance with CCDC protocol and the signed Data Use Agreement (DUA). The University of Pittsburgh Principal Investigator and study coordinator will not release any data until all request criteria are met and a signed Data Use Agreement is filed.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available beginning 6 months and ending 36 months after the primary trial results are published.
Access Criteria: All access will be thru the Center for Clinical Trials & Data Coordination (CCDC) at the University of Pittsburgh. Access will be monitored and controlled by our data center. No access will be granted until the initial requesting investigator vetting process is completed and a signed DUA is on file. All data safety plans and monitoring are listed on the CCDC website. Researchers interested in the data must sign a data use agreement (DUA) with the University of Pittsburgh, which must also be reviewed and agreed to by study partner CHASS Center Inc. No other data sharing options will be considered. The data that may be shared includes: de-identified participant data, tables, figures, appendices, analysis plan, and protocol.

REFERENCES:
- [Background] Deverts DJ, Heisler M, Kieffer EC, Piatt GA, Valbuena F, Yabes JG, Guajardo C, Ilarraza-Montalvo D, Palmisano G, Koerbel G, Rosland AM. Comparing the effectiveness of Family Support for Health Action (FAM-ACT) with traditional community health worker-led interventions to improve adult diabetes management and outcomes: study protocol for a randomized controlled trial. Trials. 2022 Oct 3;23(1):841. doi: 10.1186/s13063-022-06764-1. PMID 36192769
- [Background] Zupa MF, Perez S, Palmisano G, Kieffer EC, Piatt GA, Valbuena FM, Deverts DJ, Yabes JG, Heisler M, Rosland AM. Changes in Self-management During the COVID-19 Pandemic Among Adults with Type 2 Diabetes at a Federally Qualified Health Center. J Immigr Minor Health. 2022 Oct;24(5):1375-1378. doi: 10.1007/s10903-022-01351-7. Epub 2022 Mar 17. PMID 35301642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from a Federally Qualified Health Center (FQHC) in the mid-western US that serves a low SES, primarily Spanish-speaking population. Enrollment took place from Sep. 2019 to Dec. 2022, with a several month pause between Mar. 2020 and Feb. 2021 when restrictions were placed on in-person research. Potential participants were identified via FQHC EHR or clinician referral, and recruited by letter and phone. Support Persons were identified by patients and recruited by phone.
Pre-assignment Details: No enrolled participants were excluded before being assigned to a study arm.
Groups:
- FAM-ACT - Patients; FAM-ACT - Support Persons: FAM-ACT is a diabetes self-management education and support (DSMES) intervention for adults with type 2 diabetes ('patients') and their support persons ('SP'). The intervention consists of 3 components: an introductory session with a community health worker (CHW), 6 CHW-led DSMES sessions based on an ADA-approved DSMES curriculum, and twice-monthly care management calls. Patients and SPs are encouraged to take part in all components together. The introductory session is designed to provide an overview of diabetes complications, ways the SP and patient can work together positively, and ways to set 'SMART' health goals. During this session results of a diabetes complication risk profile are discussed with the patient and SP and the dyad learns how to set goals together. The 6 DSMES sessions last 45 minutes to 1 hour and can be conducted in person or virtually. Each topical session is enhanced with a discussion of progress toward SPs increasing their involvement in the patient's diabetes management, and skills SPs can use to address the diabetes management topics covered in the session. SP-enhanced sessions also include discussions about positive communication techniques and patient-SP weekly talks about diabetes. Patients and SPs also receive bimonthly care management calls from a CHW by phone or video chat. Calls last about 20 minutes during which the CHW discusses with the dyad the patients' progress toward their goals and ways the SP can help the patient achieve those goals.
- I-DSMES - Patients: The individual patient-focused DSMES intervention (I-DSMES) is comprised of the same 3 components described for FAM-ACT: an introductory session with a CHW, 6 CHW-led DSMES sessions based on an ADA-approved DSMES curriculum, and twice-monthly care management calls. I-DSMES differs from FAM-ACT in that the DSMES sessions are not enhanced with support-focused information and SPs are not invited to participate in the intervention with the patient. SPs in the I-DSMES arm may attend the DSMES sessions if they choose to do so, but they will not receive any SP-focused information.
- I-DSMES - Support Persons: The individual patient-focused DSMES intervention (I-DSMES) is comprised of the same 3 components described for FAM-ACT: an introductory session with a CHW, 6 CHW-led DSMES sessions based on an ADA-approved DSMES curriculum, and twice-monthly care management calls. I-DSMES differs from FAM-ACT in that the DSMES sessions are not enhanced with support-focused information and SPs are not invited to participate in the intervention with the patient. SPs in the I-DSMES arm may attend the DSMES sessions if they choose to do so, bu
Period: Baseline
Arm/Group | FAM-ACT - Patients | I-DSMES - Patients | FAM-ACT - Support Persons | I-DSMES - Support Persons
Started | 112 | 110 | 112 | 110
Completed | 112 | 110 | 112 | 110
Not Completed | 0 | 0 | 0 | 0
Period: Intervention
Arm/Group | FAM-ACT - Patients | I-DSMES - Patients | FAM-ACT - Support Persons | I-DSMES - Support Persons
Started | 112 | 110 | 112 | 110
Completed | 104 | 103 | 94 (Some Support Persons opted not to attend the introduction session with the patient, but did not formally withdraw from the study. These Support Persons still were eligible to receive their follow-up assessment.) | 22 (Support Persons in the I-DSMES arm were not invited to attend the information session. Any Support Persons who did attend did so by their own choice. Support Persons who did not attend the introduction session still were eligible to complete their follow-up assessment.)
Not Completed | 8 | 7 | 18 | 88
Not completed — Withdrawal by Subject | 7 | 2 | 7 | 2
Not completed — Patient declined to participate in the introductory session intervention | 1 | 5 | 11 | 86
Period: 6-month Follow-up
Arm/Group | FAM-ACT - Patients | I-DSMES - Patients | FAM-ACT - Support Persons | I-DSMES - Support Persons
Started | 105 (This number is greater than the number of participants who completed the intervention because any patient who actively was enrolled in the study, regardless of intervention participation, was eligible for a study A1c assessment at 6 months post-enrollment) | 108 (This number is greater than the number of participants who completed the intervention because any patient who actively was enrolled in the study, regardless of intervention participation, was eligible for a study A1c assessment at 6 months post-enrollment) | 71 (The protocol was changed after the start of the COVID-19 pandemic so that Support Persons were receiving their second assessments at 6 months rather than 12 months. The number here represents the number of FAM-ACT Support Persons who were recruited after the pandemic and so completed their follow up assessment at 6 months.) | 71 (The protocol was changed after the start of the COVID-19 pandemic so that Support Persons were receiving their second assessments at 6 months rather than 12 months. The number here represents the number of I-DSMES Support Persons who were recruited after the pandemic and so completed their follow up assessment at 6 months.)
Completed (The criterion for completing the 6-month assessment differed for patients and Support Persons. For patients, completion required having a 6-month hemoglobin A1c (A1c) value obtained either during a study visit or during a clinic visit scheduled near the time of the 6-month follow up. For Support Persons, completion of this study period was based on their completing the follow up survey assessment.) | 82 | 88 | 59 | 63
Not Completed | 23 | 20 | 12 | 8
Not completed — We were prevented from collecting A1c data from many patients due to pandemic-related restrictions | 23 | 20 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 12 | 8
Period: 12-month Follow-up
Arm/Group | FAM-ACT - Patients | I-DSMES - Patients | FAM-ACT - Support Persons | I-DSMES - Support Persons
Started | 103 (This number is greater than the number of participants who completed the 6-month assessment because any patient who actively was enrolled in the study, regardless of 6-month assessment completion, was eligible for a study A1c assessment at 12 months post-enrollment) | 108 (This number is greater than the number of participants who completed the 6-month assessment because any patient who actively was enrolled in the study, regardless of 6-month assessment completion, was eligible for a study A1c assessment at 12 months post-enrollment) | 34 (The protocol was changed after the start of the COVID-19 pandemic so that Support Persons were receiving their second assessments at 6 months rather than 12 months. The number here represents the number of FAM-ACT Support Persons who were recruited before the pandemic and so completed their follow up assessment at 12 months (less those from dyads that withdrew).) | 37 (The protocol was changed after the start of the COVID-19 pandemic so that Support Persons were receiving their second assessments at 6 months rather than 12 months. The number here represents the number of I-DSMES Support Persons who were recruited before the pandemic and so completed their follow up assessment at 12 months (less those from dyads that withdrew).)
Completed (The criterion for completing the 12-month assessment differed for patients and Support Persons. For patients, completion required having a 12-month hemoglobin A1c (A1c) value obtained either during a study visit or during a clinic visit scheduled near the time of the 12-month follow up. For Support Persons, completion of this study period was based on their completing the follow up survey assessment.) | 85 | 91 | 29 | 35
Not Completed | 18 | 17 | 5 | 2
Not completed — Lost to Follow-up | 18 | 17 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- FAM-ACT-Patients; FAM-ACT-Support Persons: Patient and Support Person (dyad) will be included together as much as possible. The dyad will:
  1. Take part in a one-hour introductory session and review of the patient's Diabetes Complications Risk Assessment profile.
  2. Be invited to 4-6 Support Person-focused, group diabetes self-management education (DSME) sessions lasting 1-2 ½ hours each.
  3. Receive case management contacts with a Community Health Worker (CHW) once every 2-4 weeks, subject to participant availability. Successful contacts will last approximately 20 minutes.
  FAM ACT: Patient and Support Person (dyad) will receive a Diabetes Complications Risk Assessment profile and introduction session, Support Person-focused information/skills training through 4-6 extended DSME sessions, case management contacts with CHW throughout the duration of the 6-month intervention, and guidance on how to prepare for and participate in healthcare appointments.
- I-DSMES-Patients: This arm will focus on the patient only. The Support Person assigned to this arm will not be invited to the introduction sessions, care management contacts, or diabetes self-management education sessions. Patients assigned to this arm will:
  1. Take part in a one-hour introductory session and review of patient's diabetes management risk assessment.
  2. Be invited to 4-6 group diabetes self-management education (DSME) sessions lasting 45 min to 2 hours each.
  3. Receive case management contacts with a Community Health Worker (CHW) once every 2-4 weeks, subject to participant availability. Successful contacts will last approximately 20 minutes.
  I-DSMES: Patient only will receive a Diabetes Complications Risk Assessment profile and introduction session, 4-6 group DSME sessions, case management contacts with CHW throughout the duration of the 6-month intervention, and guidance on how to prepare for and participate in healthcare appointments.
- I-DSMES-Support Persons: This arm will focus on the patient only. The Support Person assigned to this arm will not be invited to the introduction sessions, care management contacts, or diabetes self-management education sessions.
- Total: Total of all reporting groups
Arm/Group | FAM-ACT-Patients | I-DSMES-Patients | FAM-ACT-Support Persons | I-DSMES-Support Persons | Total
Number analyzed (Participants) | 112 | 110 | 112 | 110 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.0) | 52.8 (10.3) | 44.7 (12.7) | 46.0 (14.2) | 52.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 65 | 82 | 87 | 306
  Male | 40 | 45 | 30 | 23 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 87 | 101 | 87 | 376
  Not Hispanic or Latino | 11 | 23 | 11 | 23 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — A large proportion of participants reported "other" as their race because they identify as Latino/Hispanic for both their ethnicity and race
  Participants
    American Indian or Alaska Native | 3 | 1 | 3 | 3 | 10
    Asian | 0 | 1 | 0 | 3 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 8 | 17 | 9 | 16 | 50
    White | 8 | 14 | 16 | 15 | 53
    More than one race | 3 | 0 | 1 | 0 | 4
    Other | 90 | 77 | 83 | 73 | 323
Hemoglobin A1c (A1c) [Mean (Standard Deviation); unit: %] — The main outcome, change in A1c from baseline to 6 months, was assessed for patient participants only. Population: The main outcome, change in A1c from baseline to 6 months, was assessed for patient participants only. SP participants were not included in the analysis.
  %
    number analyzed (Participants) | 112 | 110 | 0 | 0 | 222
    (all) | 9.26 (1.85) | 9.14 (1.66) |  |  | 9.2 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient Glycemic Control at 6 Months
Description: Hemoglobin A1c (HbA1c, percent) was measured via finger stick performed by a study research assistant, by a clinician as a part of the patients' regular care, or by patients via home test kit. For analysis, HbA1c first was examined graphically to understand how it changed over time. Main analyses then were conducted using linear mixed-effects models, with 12-month HbA1c values included in the models to increase the power to estimate changes over the initial 6 months. Adjusted outcome and effect estimates at 6 months were derived from linear mixed models using linear contrasts. The model was fitted using all available time points (baseline, 6 months, and 12 months) from all 222 enrollees to make efficient use of the data. Including all time points allows the model to account for individual trajectories over time, thus increasing power to detect treatment effects and reducing bias that could arise from analyzing the 6-month time point in isolation.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete HbA1c data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: percentage
Groups:
- FAM-ACT: FAM-ACT is a diabetes self-management education and support (DSMES) intervention for adults with type 2 diabetes ('patients') and their support persons ('SP'). The intervention consists of 3 components: an introductory session with a community health worker (CHW), 6 CHW-led DSMES sessions based on an ADA-approved DSMES curriculum, and twice-monthly care management calls. Patients and SPs are encouraged to take part in all components together. The introductory session is designed to provide an overview of diabetes complications, ways the SP and patient can work together positively, and ways to set 'SMART' health goals. During this session results of a diabetes complication risk profile are discussed with the patient and SP and the dyad learns how to set goals together. The 6 DSMES sessions last 45 minutes to 1 hour and can be conducted in person or virtually. Each topical session is enhanced with a discussion of progress toward SPs increasing their involvement in the patient's diabetes management, and skills SPs can use to address the diabetes management topics covered in the session. SP-enhanced sessions also include discussions about positive communication techniques and patient-SP weekly talks about diabetes. Patients and SPs also receive bimonthly care management calls from a CHW by phone or video chat. Calls last about 20 minutes during which the CHW discusses with the dyad the patients' progress toward their goals and ways the SP can help the patient achieve those goals.
- I-DSMES: The individual patient-focused DSMES intervention (I-DSMES) is comprised of the same 3 components described for FAM-ACT: an introductory session with a CHW, 6 CHW-led DSMES sessions based on an ADA-approved DSMES curriculum, and twice-monthly care management calls. I-DSMES differs from FAM-ACT in that the DSMES sessions are not enhanced with support-focused information and SPs are not invited to participate in the intervention with the patient. SPs in the I-DSMES arm may attend the DSMES sessions if they choose to do so, but they will not receive any SP-focused information.
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 82 | 88
percentage | -0.43 [-0.85 to -0.00] | -0.97 [-1.38 to -0.55]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Linear mixed model with random intercept and slope was used to compare the change in HbA1c as a function of time (included using restricted cubic splines), the interaction between time and intervention arm, baseline A1c and whether PT-SP live together (stratification variables), baseline insulin use, age, vital hunger, and preferred language; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [-0.05 to 1.14] — Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

2. Secondary Outcome: Change From Baseline in Patient Glycemic Control at 12 Months
Description: Hemoglobin A1c (HbA1c, percent) was measured through finger stick performed by a study research assistant, by a clinician as a part of the patients' regular care, or by the patients themselves via a home test kit.
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete HbA1c data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: percentage
Groups:
- FAM-ACT: Patient and Support Person (dyad) will be included together as much as possible. The dyad will:
  1. Take part in a one-hour introductory session and review of the patient's Diabetes Complications Risk Assessment profile.
  2. Be invited to 4-6 Support Person-focused, group diabetes self-management education (DSME) sessions lasting 1-2 ½ hours each.
  3. Receive case management contacts with a Community Health Worker (CHW) once every 2-4 weeks, subject to participant availability. Successful contacts will last approximately 20 minutes.
  FAM ACT: Patient and Support Person (dyad) will receive a Diabetes Complications Risk Assessment profile and introduction session, Support Person-focused information/skills training through 4-6 extended DSME sessions, case management contacts with CHW throughout the duration of the 6-month intervention, and guidance on how to prepare for and participate in healthcare appointments.
- I-DSMES: This arm will focus on the patient only. The Support Person assigned to this arm will not be invited to the introduction sessions, care management contacts, or diabetes self-management education sessions. Patients assigned to this arm will:
  1. Take part in a one-hour introductory session and review of patient's diabetes management risk assessment.
  2. Be invited to 4-6 group diabetes self-management education (DSME) sessions lasting 45 min to 2 hours each.
  3. Receive case management contacts with a Community Health Worker (CHW) once every 2-4 weeks, subject to participant availability. Successful contacts will last approximately 20 minutes.
  I-DSMES: Patient only will receive a Diabetes Complications Risk Assessment profile and introduction session, 4-6 group DSME sessions, case management contacts with CHW throughout the duration of the 6-month intervention, and guidance on how to prepare for and participate in healthcare appointments.
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 85 | 91
percentage | -0.67 [-1.14 to -0.20] | -0.65 [-1.11 to -0.19]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Linear mixed model with random intercept and slope was used to compare the change in A1c as a function of time (included using restricted cubic splines), the interaction between time and intervention arm, baseline A1c and whether PT-SP live together (stratification variables), baseline insulin use, age, vital hunger, and preferred language; Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.67 to 0.64] — Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

3. Secondary Outcome: Change From Baseline in Patient Systolic Blood Pressure at 6 Months
Description: SBP was measured using an electronic, upper arm blood pressure monitor.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete SBP data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 82 | 86
mmHg | -0.85 [-4.33 to 2.63] | 0.66 [-2.78 to 4.10]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient SBP was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.55, Mixed Models Analysis; Mean Difference (Final Values) = -1.51, 95% CI 2-sided [-6.40 to 3.38] — Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

4. Secondary Outcome: Change From Baseline in Patient Systolic Blood Pressure at 12 Months
Description: SBP was measured using an electronic, upper arm blood pressure monitor.
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete SBP data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 79 | 87
mmHg | 2.69 [-0.98 to 6.35] | -3.05 [-6.70 to 0.59]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = 5.74, 95% CI 2-sided [0.57 to 10.91] — Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

5. Secondary Outcome: Change From Baseline in Patient Diabetes Distress at 6 Months
Description: Patient diabetes distress was assessed using the Problem Areas in Diabetes (PAID-5) Scale. The scale is comprised of 5 closed-ended items with response options ranging from 0 ('not a problem') to 4 ('serious problem'). The scale's 5 items were summed to create a total score with a range of 0 to 20. A total score of >=8 indicates possible diabetes-related emotional distress that warrants further assessment, with higher scores suggesting greater diabetes-related emotional distress.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete PAID-5 data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 93 | 101
score on a scale | -2.68 [-4.01 to -1.35] | -2.40 [-3.71 to -1.09]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient diabetes distress was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.76, Mixed Models Analysis; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-2.15 to 1.58] — Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

6. Secondary Outcome: Change From Baseline in Patient Diabetes Distress at 12 Months
Description: as for outcome 5
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete PAID-5 data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 84 | 96
score on a scale | -2.67 [-3.94 to -1.39] | -2.34 [-3.59 to -1.10]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-2.11 to 1.46] — Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

7. Secondary Outcome: Change From Baseline Patient Diabetes Self-care Behaviors at 6 Months: Healthy Eating
Description: The Summary of Diabetes Self-Care Activities (SDSCA) is a brief self-report instrument for measuring levels of self-management across different components of the diabetes regimen. Results were scored separately within each domain. Scores range from 1 to 7, representing the number of days per week the patient engages in the behavior. Higher numbers indicate better adherence.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete SDSCA diet data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 93 | 101
score on a scale | 0.14 [-0.24 to 0.51] | 0.37 [-0.00 to 0.74]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient health eating was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.38, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.76 to 0.29] — Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

8. Secondary Outcome: Change in Diabetes Self-care Behaviors in Patient: Physical Activity
Description: as for outcome 7
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete SDSCA physical activity data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 93 | 101
units on a scale | 0.52 [-0.14 to 1.17] | 0.70 [0.05 to 1.35]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient physical activity was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-1.11 to 0.74] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

9. Secondary Outcome: Change in Diabetes Self-care Behaviors in Patient: Medication Adherence
Description: The Summary of Diabetes Self-Care Activities (SDSCA) is a brief self-report instrument for measuring levels of self-management across different components of the diabetes regimen. Results were scored separately within each domain. Scores range from 1 to 7, representing the number of days per week the patient engages in the behavior. Higher numbers indicate better adherence. Three types of medication adherence were assessed: number of days diabetes medications (non-insulin) were taken; number of days blood pressure medications were taken; number of days cholesterol medications were taken. Note that the Ns with data for these three measures are smaller than the Ns for diet and physical activity data. Differences are due to some patients not having been prescribed non-insulin diabetes, blood pressure and/or cholesterol medications.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 patient participants enrolled in the study. Ns represent the number of adult patients with type 2 diabetes who had complete adherence data for diabetes, blood pressure, and cholesterol medications, respectively, at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 85 | 93
units on a scale
  Diabetes medication | 0.12 [-0.34 to 0.58] | 0.01 [-0.43 to 0.45]
  Blood pressure medication: number analyzed (Participants) | 59 | 49
  Blood pressure medication | 0.05 [-0.56 to 0.66] | 0.09 [-0.64 to 0.81]
  Cholesterol medication: number analyzed (Participants) | 53 | 46
  Cholesterol medication | 0.01 [-0.69 to 71] | 0.44 [-0.32 to 1.20]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient diabetes medication adherence was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.75, Mixed Models Analysis; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.53 to 0.74] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES
Statistical Analysis 2: Comparison: FAM-ACT vs I-DSMES; Change in patient blood pressure medication adherence (days/week meds were taken) was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c). Analyses were ITT and thus based on data from all enrolled patients; Test type: Superiority; p = 0.94, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.98 to 0.91] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES
Statistical Analysis 3: Comparison: FAM-ACT vs I-DSMES; Change in patient cholesterol medication adherence (days/week meds were taken) was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c). Analyses were ITT and thus based on data from all enrolled patients; Test type: Superiority; p = 0.42, Mixed Models Analysis; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.46 to 0.61] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

10. Secondary Outcome: Change in Self-efficacy of Patient
Description: Patient self-efficacy for managing diabetes was assessed with the Self-Efficacy for Managing Chronic Diseases Scale. The scale is comprised of 5 items asking respondents to indicate how confident they are that they regularly can perform tasks related to their diabetes management (0, not at all confident to 10, very confident). Item responses are averaged, with mean scores ranging from 0 to 10. Higher numbers indicate greater self-efficacy.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete self-efficacy data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 93 | 101
units on a scale | 0.33 [-0.05 to 0.71] | 0.34 [-0.03 to 0.72]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient self-efficacy was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.54 to 0.52] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

11. Secondary Outcome: Change in Patient Activation in Patient
Description: Patient activation was assessed with the Patient Activation Measure (PAM)-10. Using a 4-point scale (1=strongly disagree to 4=strongly agree), respondents indicate the extent to which statements related to being ready, willing and able to manage their health and health care accurately describe them. Responses are summed to create a total score with higher numbers indicating greater activation. Item scale locations were transformed from the original logit metric to a user-friendly 0-100 metric where 0=the lowest possible activation and 100=the highest possible activation as measured by this set of items. While the metric allows for a potential range of 0-100, the items included in the measure only covered the range from 40 (minimum) to 60 (maximum), not tapping what would be theoretically the lowest or highest ranges of the construct.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete patient activation data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 93 | 101
units on a scale | 5.95 [1.08 to 10.82] | 3.02 [-1.79 to 7.84]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient activation was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.40, Mixed Models Analysis; Mean Difference (Final Values) = 2.93, 95% CI 2-sided [-3.92 to 9.78] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

12. Secondary Outcome: Patient Perceived Overall Satisfaction With SP Support for Diabetes
Description: Patient satisfaction with support person (SP) support for diabetes was assessed with 2* items assessing patient's satisfaction with the support they receive from their SP and whether they feel like they would be worse off without their SP's help with their diabetes care. Responses were rated on a 7-point scale ranging from 1, "strongly disagree" to 7 "strongly agree". Responses are summed to create a total score with a range of 2 to 14. Higher numbers indicate greater satisfaction.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete support satisfaction data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 93 | 100
units on a scale | 0.38 [-0.29 to 1.04] | -0.37 [-1.03 to 0.28]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient satisfaction with SP support was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Final Values) = 0.75, 95% CI 2-sided [-0.18 to 1.68] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

13. Secondary Outcome: Patient Perception of SP Support: Supportive and Non-supportive Behaviors
Description: Patient perception of support persons' (SP) supportive behaviors was assessed using the 8-item Important Other Climate Questionnaire (IOCQ) and non-supportive behaviors using 3 similarly-structured items addressing SP irritation, criticism and argumentativeness. All items are rated on a 7-point scale ranging from 0 ("strongly disagree") to 6 ("strongly agree"), with non-supportive behavior items being reversed scored. Item responses were averaged to create a mean score with a possible range of 0 (low support) to 6 (high support).
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete IOCQ data at both baseline and 6-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 93 | 101
units on a scale | 0.22 [-0.04 to 0.49] | 0.04 [-0.22 to 0.30]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient perception of supportive and non-supportive behaviors was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.34, Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.19 to 0.55] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

14. Secondary Outcome: Impact of COVID on Ability to Manage Diabetes
Description: Impact of COVID on ability to manage Diabetes was assessed with a single closed-ended item: "In the last six months, how have the COVID pandemic or social distancing rules affected your ability to manage your diabetes?" The item is rated on a 5-point scale ranging from "much harder" to "much easier". Due to small numbers, the variable was collapsed to 3 categories for analysis: harder/much harder, no change, easier/much easier.
Time Frame: Cross-sectional at 6 months
Population: All patient participants with complete impact of COVID on diabetes management data.
Measure: Count of Participants; unit: Participants
Arm/Group | FAM-ACT - Patients | I-DSMES - Patients
Number analyzed (Participants) | 61 | 69
Participants
  Harder/much harder | 6 | 4
  No change | 53 | 64
  Easier/much easier | 2 | 1

15. Secondary Outcome: Change in Diabetes Distress in Support Person
Description: Support person distress about the patient's diabetes was assessed using the Problem Areas in Diabetes (PAID-5) Scale (for family members). The scale is comprised of 5 closed-ended items with response options ranging from 0 ('not a problem') to 4 ('serious problem'). The scale's 5 items were summed to create a total score with a range of 0 to 20. A total score of >=8 indicates possible diabetes-related emotional distress that warrants further assessment, with higher scores suggesting greater diabetes-related emotional distress.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 support persons enrolled in the study. Ns represent the number of support persons who had complete PAID-5 data at both baseline and 6-months post-baseline. See comments on Statistical Analysis 1 for additional detail.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 59 | 63
units on a scale | -1.99 [-3.35 to -0.63] | -1.27 [-2.67 to 0.12]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Support Persons (SPs) were surveyed twice, once at baseline and again at the end of their participation in the study. For SPs enrolled before the start of the COVID-19 pandemic (n=77), the follow-up survey was conducted at 12 months. Due to factors related to the pandemic, the length of the protocol was reduced from 12 to 6 months. Thus, SPs enrolled after the pandemic started (n=145) received their follow-up survey at 6 months, and 6-month change was used for predetermined SP outcomes; Test type: Superiority; p = 0.47, Mixed Models Analysis; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-2.67 to 1.23] — Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

16. Secondary Outcome: Change in Self-efficacy of Support Person
Description: Support person self-efficacy for helping the patient with managing diabetes was assessed with the Self-Efficacy for Managing Chronic Diseases Scale (adapted for support persons). The scale is comprised of 5 items asking respondents to indicate how confident they are that they regularly can help patients perform tasks related to their diabetes management (0, not at all confident to 10, very confident). Item responses are averaged, with mean scores ranging from 0 to 10. Higher numbers indicate greater self-efficacy.
Time Frame: Baseline vs. 6 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 support persons enrolled in the study. Ns represent the number of support persons who had complete self-efficacy data at both baseline and 6-months post-baseline. See comments on Statistical Analysis 1 for additional detail.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 59 | 63
units on a scale | -0.27 [-0.64 to 0.10] | -0.02 [-0.39 to 0.36]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.35, Mixed Models Analysis; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.78 to 0.27] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

17. Other Pre Specified Outcome: Change in Diabetes Self-care Behaviors in Patient: Healthy Eating
Description: as for outcome 7
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete SDSCA diet data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 84 | 96
units on a scale | -0.09 [-0.45 to 0.27] | 0.41 [0.05 to 0.76]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Change in patient healthy eating was analyzed in a manner similar to that described for the primary outcome (6-month change in patient A1c); Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.00 to 0.01] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

18. Other Pre Specified Outcome: Change in Diabetes Self-care Behaviors in Patient: Physical Activity
Description: as for outcome 7
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete SDSCA physical activity data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 84 | 96
units on a scale | 0.22 [-0.41 to 0.85] | 0.56 [-0.06 to 1.17]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Test type: Superiority; p = 0.45, Mixed Models Analysis; Median Difference (Final Values) = -0.34, 95% CI 2-sided [-1.22 to 0.54] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

19. Other Pre Specified Outcome: Change in Diabetes Self-care Behaviors in Patient: Medication Adherence
Description: The Summary of Diabetes Self-Care Activities (SDSCA) is a brief self-report instrument for measuring levels of self-management across different components of the diabetes regimen. Results were scored separately within each domain. Scores range from 1 to 7, representing the number of days per week the patient engages in the behavior. Higher numbers indicate better adherence. Three types of medication adherence were assessed: number of days diabetes medications (non-insulin) were taken; number of days blood pressure medications were taken; number of days cholesterol medications were taken. Note that the Ns with data for these three measures are smaller than the Ns for diet and physical activity data. Differences are due to patients not having been prescribed non-insulin diabetes, blood pressure and/or cholesterol medications.
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete adherence data for diabetes, blood pressure, and cholesterol medication, respectively, at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT-Patients | I-DSMES-Patients
Number analyzed (Participants) | 76 | 88
units on a scale
  Diabetes medications | 0.01 [-0.42 to 0.44] | 0.27 [-0.16 to 0.69]
  Blood pressure medications: number analyzed (Participants) | 51 | 46
  Blood pressure medications | 0.04 [-0.57 to 0.65] | 0.05 [-0.60 to 0.70]
  Cholesterol medications: number analyzed (Participants) | 47 | 88
  Cholesterol medications | -0.02 [-0.72 to 0.68] | 0.39 [-0.34 to 1.12]
Statistical Analysis 1: Comparison: FAM-ACT-Patients vs I-DSMES-Patients; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.40, Mixed Models Analysis; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.86 to 0.35] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES
Statistical Analysis 2: Comparison: FAM-ACT-Patients vs I-DSMES-Patients; Change in patient blood pressure medication adherence (days/week meds were taken) was analyzed in a manner similar to that described for the primary outcome (6month change in patient A1c). Analyses were ITT and thus based on data from all enrolled patients; Test type: Superiority; p = 0.98, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.90 to 0.88] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES
Statistical Analysis 3: Comparison: FAM-ACT-Patients vs I-DSMES-Patients; Change in patient cholesterol medication adherence (days/week meds were taken) was analyzed in a manner similar to that described for the primary outcome (6month change in patient A1c). Analyses were ITT and thus based on data from all enrolled patients; Test type: Superiority; p = 0.43, Mixed Models Analysis; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-1.42 to 0.61] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

20. Other Pre Specified Outcome: Change in Self-efficacy of Patient
Description: as for outcome 10
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete self-efficacy data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 84 | 96
units on a scale | 0.09 [-0.27 to 0.46] | 0.59 [0.23 to 0.94]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.00 to 0.01] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

21. Other Pre Specified Outcome: Change in Patient Activation in Patient
Description: as for outcome 11
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete patient activation data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 84 | 96
units on a scale | 3.18 [-1.72 to 8.08] | 3.54 [-1.24 to 8.33]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.92, Mixed Models Analysis; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-7.22 to 6.49] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

22. Other Pre Specified Outcome: Patient Perceived Overall Satisfaction With Support Person Support for Diabetes
Description: as for outcome 12
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete support satisfaction data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 82 | 95
units on a scale | 0.55 [-0.09 to 1.19] | -0.55 [-1.17 to 0.07]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = 1.10, 95% CI 2-sided [0.21 to 1.99] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

23. Other Pre Specified Outcome: Patient Perception of Support Person Support: Supportive and Non-supportive Behaviors
Description: as for outcome 13
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete IOCQ data at both baseline and 12-months post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT - Patients | I-DSMES - Patients
Number analyzed (Participants) | 82 | 96
units on a scale | 0.30 [0.05 to 0.56] | -0.04 [-0.29 to 0.21]
Statistical Analysis 1: Comparison: FAM-ACT - Patients vs I-DSMES - Patients; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.01 to 0.70] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

24. Other Pre Specified Outcome: Change in Diabetes Distress in Support Person
Description: as for outcome 15
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 support persons enrolled in the study. Ns represent the number of enrolled support persons who had complete PAID-5 data at both baseline and 12-months post-baseline. See comments on Statistical Analysis 1 for additional detail.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 29 | 35
units on a scale | 0.45 [-1.99 to 2.90] | -0.74 [-3.07 to 1.60]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.49, Mixed Models Analysis; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-2.19 to 4.57]; Positive coefficient favors I-DSMES; negative coefficient favors FAM-ACT

25. Other Pre Specified Outcome: Change in Self-efficacy of Support Person
Description: as for outcome 16
Time Frame: Baseline vs. 12 months
Population: Analyses were Intention-to-Treat (ITT) and thus were based on data from all 222 adults with type 2 diabetes enrolled in the study. Ns represent the number of enrolled adults with type 2 diabetes who had complete self-efficacy data at both baseline and 12-months post-baseline.See comments on Statistical Analysis 1 for additional detail.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | FAM-ACT | I-DSMES
Number analyzed (Participants) | 29 | 35
units on a scale | 0.07 [-0.57 to 0.70] | -0.72 [-1.32 to -0.11]
Statistical Analysis 1: Comparison: FAM-ACT vs I-DSMES; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = 0.78, 95% CI 2-sided [-0.09 to 1.66] — Positive coefficient favors FAM-ACT; negative coefficient favors I-DSMES

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 1 year, beginning at the time of randomization and ending after the 12-month study assessment.
Description: Study staff were trained to report all AEs and potential problems immediately. Also, the informed consent document contained contact information for the PI and University of Pittsburgh IRB to facilitate self-report of AEs. SAEs were to be categorized by the study monitor according to the CTCAE. The PI or Site-PI were responsible for adjudicating all SAEs with the aid of discharge summaries.
Groups:
- I-DSMES-Support Persons: This arm will focus on the patient only. The Support Person assigned to this arm will not be invited to the introduction sessions, care management contacts, or diabetes self-management education sessions. Patients assigned to this arm will:
  1. Take part in a one-hour introductory session and review of patient's diabetes management risk assessment.
  2. Be invited to 4-6 group diabetes self-management education (DSME) sessions lasting 45 min to 2 hours each.
  3. Receive case management contacts with a Community Health Worker (CHW) once every 2-4 weeks, subject to participant availability. Successful contacts will last approximately 20 minutes.
  I-DSMES: Patient only will receive a Diabetes Complications Risk Assessment profile and introduction session, 4-6 group DSME sessions, case management contacts with CHW throughout the duration of the 6-month intervention, and guidance on how to prepare for and participate in healthcare appointments.
Arm/Group | FAM-ACT-Patients | I-DSMES-Patients | FAM-ACT-Support Persons | I-DSMES-Support Persons
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/110 | 0/112 | 0/110
Serious Adverse Events (participants affected / at risk) | 18/112 | 20/110 | 0/112 | 0/110
Other Adverse Events (participants affected / at risk) | 38/112 | 31/110 | 0/112 | 0/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAM-ACT-Patients (N=112) | I-DSMES-Patients (N=110) | FAM-ACT-Support Persons (N=112) | I-DSMES-Support Persons (N=110)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA | NA — Abdominal pain and/or vomiting requiring hospital admission. Unrelated to study participation.
Blood clot (Vascular disorders) | 1 (1) | 0 (0) | NA | NA — Blood clot requiring hospital admission. Unrelated to study participation.
Pulmonary emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | NA | NA — Pulmonary emphysema exacerbation requiring hospital admission. Unrelated to study participation.
Kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1) | NA | NA — Kidney pain requiring hospital admission. Unrelated to study participation.
COVID-19 complications (Infections and infestations) | 2 (2) | 0 (0) | NA | NA — COVID-19 complications requiring hospital admission. Unrelated to study participation.
Hospital admission, unspecified (General disorders) | 14 (14) | 17 (17) | NA | NA — Hospital admission unrelated to study participation with no additional information.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAM-ACT-Patients (N=112) | I-DSMES-Patients (N=110) | FAM-ACT-Support Persons (N=112) | I-DSMES-Support Persons (N=110)
COVID-19 (Infections and infestations) | 8 (10) | 7 (7) | NA | NA — Tested positive for COVID-19. Unrelated to study participation.
Injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | NA | NA — Patient 1, finger laceration; patient 2, foot laceration; patient 3, puncture wound to foot; patient 4, fall. All resulted in a visit to a hospital emergency department without inpatient admission. None related to study participation.
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA — Shortness of breath resulting in a visit to a hospital emergency department. No inpatient admission. Unrelated to study participation.
Fibromyalgia pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | NA | NA — Exacerbation of existing fibromyalgia pain resulting in a visit to a hospital emergency department. No inpatient admission. Unrelated to study participation.
Emergency department, unspecified (General disorders) | 25 (52) | 23 (35) | NA | NA — Unspecified events resulting in a visit to a hospital emergency department without inpatient admission. Unrelated to study participation.

LIMITATIONS AND CAVEATS:
Many patients were due for the 6-month A1c measure (main outcome) during the height of the COVID-19 pandemic when restrictions on face-to-face research activities prevented us from collecting the data and they missed this outcome window. Two compensatory strategies were enacted: (a) review patients' EHR to identify additional A1c data during the collection window and (b) send patients home A1c test kits. This did yield some additional data, but we still missed 6-month A1c data for many patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT03812614/Prot_001.pdf
  • Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT03812614/SAP_002.pdf
  • Informed Consent Form (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT03812614/ICF_000.pdf